CLINICAL TRIAL: NCT00627172
Title: Combined Use of Coronary MDCTA, Coronary Doppler Ultrasonography and PET Perfusion in Diagnosis of Coronary Artery Disease
Brief Title: Combined Use of Coronary MDCTA, Coronary Doppler Ultrasonography and PET Perfusion in Diagnosing Coronary Artery Disease
Acronym: PECTUS
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Juhani Knuuti, Director, Turku PET Centre
Other Study IDs: 15559
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; MDCT; Positron emission tomography; Ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Multislice CT angiography is a novel but already established and widely used in diagnosing coronary artery disease (CAD). It is very reliable in ruling out hemodynamically significant narrowings in coronary arteries (Negative predictive value). However, it may overestimate the severity of the stenoses in up to 30% of the coronary artery lesions (positive predictive value 70%). However, when coupled with a functional or flow-sensitive diagnostic test, such as PET perfusion or coronary doppler ultrasonography, one can assume that even the PPV may be as high as 95 %. Despite this assumption, there's no scientific evidence to support use of such hybrid multi-modality tests at present.

The investigators hypothesis is that improving the diagnostic accuracy of non-invasive diagnosis of coronary artery disease will decrease the proportion of patients that need catheter angiographies. The avoidance of these unnecessary invasive procedures will improve patients´ quality of life and may even redirect health care resources in a more efficient way.

DETAILED DESCRIPTION:
Coronary MDCTA (multi-detector CT angiography) is a novel but already established and widespread diagnostic method to diagnose coronary artery disease. When performed with a 64-detector (slice) CT, its strength is an excellent negative predictive value, NPV (98%). Specificity (86%) is good but the positive predictive value (PPV) is only moderate (70%). This is due to the ability of MDCTA to detect even minor vessel wall changes before they are functionally significant, and the tendency of CT to overestimate the volume of dense calcifications. However, when coupled with a functional or flow-sensitive diagnostic test, such as PET perfusion or coronary doppler ultrasonography, one can assume that even the PPV may be as high as 95 %. Despite this assumption, there's no scientific evidence to support use of such hybrid multi-modality tests at present.

Our hypothesis is that improving the diagnostic accuracy of non-invasive diagnosis of coronary artery disease will decrease the proportion of patients that need catheter angiographies. The avoidance of these unnecessary invasive procedures will improve patients´ quality of life and may even redirect health care resources in a more efficient way.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age 40 - 80 years
* stable chest pain
* likelihood of obstructive coronary artery disease more than 25% based on gender, age, symptoms and exercise test

Exclusion Criteria:

* irregular rhythm
* hypersensitivity to contrast agents
* unstable chest pain
* decompensated congestive heart failure
* abnormal kidney function
* 2nd or 3rd degree AV block
* severe bronchial asthma
* pregnancy
* age over 80 years
* previously diagnosed coronary artery disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-01; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Detection of hemodynamically significant coronary artery lesions with combined use coronary CT and PET perfusion as compared with invasive angiography combined with measurement of fractional flow reserve | In the beginning of the study

SECONDARY OUTCOMES:
Detection of hemodynamically significant coronary artery lesions with combined use coronary CT and coronary doppler ultrasonography as compared with invasive angiography combined with measurement of fractional flow reserve | In the beginning of the study
Quality of life | Baseline and at 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Turku PET Centre, Turku
  - Turku University Hospital, Department of Medicine, Turku

REFERENCES:
- [Derived] Kajander SA, Joutsiniemi E, Saraste M, Pietila M, Ukkonen H, Saraste A, Sipila HT, Teras M, Maki M, Airaksinen J, Hartiala J, Knuuti J. Clinical value of absolute quantification of myocardial perfusion with (15)O-water in coronary artery disease. Circ Cardiovasc Imaging. 2011 Nov;4(6):678-84. doi: 10.1161/CIRCIMAGING.110.960732. Epub 2011 Sep 16. PMID 21926262
- [Derived] Bucci M, Joutsiniemi E, Saraste A, Kajander S, Ukkonen H, Saraste M, Pietila M, Sipila HT, Teras M, Maki M, Airaksinen KE, Hartiala J, Knuuti J, Iozzo P. Intrapericardial, but not extrapericardial, fat is an independent predictor of impaired hyperemic coronary perfusion in coronary artery disease. Arterioscler Thromb Vasc Biol. 2011 Jan;31(1):211-8. doi: 10.1161/ATVBAHA.110.213827. Epub 2010 Oct 28. PMID 21030717
- [Derived] Kajander S, Joutsiniemi E, Saraste M, Pietila M, Ukkonen H, Saraste A, Sipila HT, Teras M, Maki M, Airaksinen J, Hartiala J, Knuuti J. Cardiac positron emission tomography/computed tomography imaging accurately detects anatomically and functionally significant coronary artery disease. Circulation. 2010 Aug 10;122(6):603-13. doi: 10.1161/CIRCULATIONAHA.109.915009. Epub 2010 Jul 26. PMID 20660808